CLINICAL TRIAL: NCT04918823
Title: Novel Use of Restasis (Cyclosporine Ophthalmic Emulsion 0.05%) on Application of PROSE Devices for Management of Patients With Ocular Surface Disease: A Pilot Study
Brief Title: Novel Use of Cyclosporine Ophthalmic Emulsion 0.05% in a PROSE Device
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Sight (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Daniel C Brocks, Chief Medical Officer, Boston Sight
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFS-REGEN-01
Record Dates: First submitted 2021-05-28; First posted 2021-06-09 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Ocular Surface Disease
Keywords: ocular surface disease; Restasis
MeSH Terms: interventions — Cyclosporins

STUDY DESIGN:
Intervention Model Description: All subjects will receive study drug to be used in their device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm (Other): All subjects will receive Restasis in this study
  Interventions: Drug: Restasis

INTERVENTIONS:
Drug: Restasis — Subject will use one drop of Restasis in the lens before insertion
  Other Names: cyclosporine ophthalmic solution 0.05%

SUMMARY:
The goal of this prospective observational pilot study is to evaluate the tolerability and safety of RESTASIS (cyclosporine ophthalmic solution 0.05%) when added to the PROSE (Prosthetic Replacement of the Ocular Surface Ecosystem) lens reservoir in patients with ocular surface disease (OSD). Secondary endpoints include early (1-month) efficacy data for ocular signs and symptoms.

DETAILED DESCRIPTION:
For this study, all subjects will receive Restasis (Cyclosporine ophthalmic emulsion 0.05%). One drop of the dispensed study drop will be instilled in the PROSE lens reservoir twice a day and the remainder of the reservoir will be filled with normal saline (0.9% sodium chloride solution). In order to standardize solutions used in the PROSE reservoir, all patients recruited will be either currently using or will be switched to buffered preservative-free normal saline (Purilens, Lifestyle Inc., pH 7.46 ) to better match the reported pH of RESTASIS (pH 6.5-8.05 ).

Outcomes will include subjective responses regarding the subject's symptoms and visual function in addition to the objective assessments of the health of the ocular surface seen on clinical examination. Results will be measured at baseline, after 1 week, and after 1 month of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent has been obtained prior to any study-related procedures taking place
2. Subject is Male or Female, 18 years of age or older prior to the initial visit
3. Is an established wearer of PROSE devices for > 6 months in both eyes
4. Has a finalized PROSE lens design in both eyes, in the opinion of the clinician
5. The PROSE design does NOT include fenestrations
6. Subject requires PROSE devices to treat symptoms and/or signs from underlying dry eye disease, GVHD, Sjogren's syndrome, limbal stem cell deficiency, keratoconjunctivitis sicca, or ocular surface disease
7. Baseline Corneal staining grade of 2 or higher in total, both eyes combined (NEI Grading System) 7
8. Baseline Ocular Surface Disease Index 13 or greater
9. In the opinion of the investigator, the subject can follow study instructions
10. In the opinion of the investigator, the subject can complete all study procedures and visits
11. Able to wear PROSE device continuously for at least 6 hours at a time without removal, in each eye
12. Able to wear PROSE device for at least 10 total hours a day, in each eye
13. Able to wear PROSE device in subsequent continuous sessions of 6 hours, followed by a break to re-instill Restasis in device bowl, followed by another period of continuous wear of at least 4 hours
14. Currently using buffered preservative free normal saline (Purilens) in the device bowl or willing to transition to buffered preservative free normal saline (Purilens) use in the device bowl during the study

Exclusion Criteria:

1. Is currently participating in any other type of eye-related clinical or research study
2. Is pregnant or nursing as reported by the subject.
3. Has a condition or is in a situation which, in the investigator's opinion, may put the subject at significant risk, may confound study outcomes, or may significantly interfere with the subject's participation in the study.
4. Has had previous ocular surgery within the past 12 weeks.
5. Currently uses or has a prior history of using Restasis in the last 3 months
6. Currently uses or has a prior history of using Cequa in the last 3 months
7. Is currently using Xiidra and has been using Xiidra for less than 3 months
8. Has a history of an allergic reaction or hypersensitivity to any active or inactive ingredient found in Restasis or Cequa or Purilens.
9. Is wearing a PROSE device with Tangible HydraPEG coating
10. The subject is not wearing their PROSE devices daily
11. The subject is only wearing a device for one eye.
12. The participant is monocular
13. The subject wears a PROSE lens with fenestrations
14. The participant carries a diagnosis of glaucoma or ocular hypertension or glaucoma suspect AND is currently using glaucoma medications
15. The participant is NOT able to wear PROSE devices for 6 hours continuously, followed by a break to re-instill Restasis, followed by an additional period of at least 4 hours of continuous wear
16. Allergy to sodium fluorescein
17. Allergy to lissamine green
18. Allergy or intolerance to Purilens solution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Brocks, MD, Principal Investigator — Boston Sight
Locations (1):
- BostonSight, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no IPD

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 54.3 [38 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9
Dry eye [Number; unit: participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Disease Index (OSDI) Score Change (1 Month Post Treatment Initiation)
Description: The Ocular Surface Disease Index (OSDI) is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease.
Time Frame: 1 month post initiation change in OSDI score
Population: Subjects who completed the study
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 9
score on a scale | -3.83 (6.87)

2. Primary Outcome: Corneal Staining
Description: Corneal fluorescein staining, pre and post initiation of 0.05% cyclosporine treatment, is measured using the National Eye Institute (NEI) grading system. The NEI grading scale is a system for grading corneal fluorescein staining which divides the corneal surface into 5 areas [central, superior, nasal, inferior, temporal]. A standardized grading system of 0 to 3, with 0 being no staining (better outcome) and 3 being severe staining (worse outcome), is used for each of the areas of cornea. The scores from each corneal area are totaled to determine the total corneal staining score in each eye. The total corneal staining score has a minimum score of zero (better outcome) and a maximum score of 15 (worse outcome) for an individual eye.
Time Frame: at baseline and at 1-month post treatment initiation
Population: Subjects who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 9
Number analyzed (eyes) | 18
score on a scale
  Baseline corneal staining (NEI grading system) | 11.89 (5.11)
  1-month post treatment initiation corneal staining (NEI grading system) | 5.22 (4.49)

3. Primary Outcome: Conjunctival Staining
Description: Conjunctival fluorescein staining, pre and post initiation of 0.05% cyclosporine treatment, is measured using the National Eye Institute (NEI) grading system. The NEI grading scale is a system for grading conjunctival fluorescein staining which divides the conjunctival surface into 6 areas. A standardized grading system of 0 to 3, with 0 being no staining (better outcome) and 3 being severe staining (worse outcome), is used for each of the areas of conjunctiva. The scores from each conjunctival area are totaled to determine the total conjunctival staining score in each eye. The total conjunctival staining score has a minimum score of zero (better outcome) and a maximum score of 18 (worse outcome) for an individual eye.
Time Frame: baseline and 1-month post treatment initiation
Population: Subjects who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 9
Number analyzed (eyes) | 18
score on a scale
  Conjunctival staining (NEI grading system) at baseline | 12.22 (10.49)
  Conjunctival staining (NEI grading system) at 1-month post treatment initiation | 7.11 (7.74)

4. Primary Outcome: Visual Acuity
Description: Subjects vision was tested using Snellen visual acuity chart (converted to LogMAR scale) pre and post initiation of 0.05% cyclosporine treatment. The LogMAR scale ranges from +3.00 to -0.30. A Zero LogMAR indicates standard 20/20 vision. More negative logMAR scale vision indicates better vision. More positive logMAR scale vision indicates worse vision. Legal blindness is defined as a best-corrected visual acuity of +1.0 LogMAR pr worse in the better seeing eye.
Time Frame: at baseline and 1-month post treatment initiation
Population: Subjects who completed the study
Measure: Mean (Standard Deviation); unit: score on a logMAR scale
Units Other Than Participants: eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 9
Number analyzed (eyes) | 18
score on a logMAR scale
  BCVA baseline | 0.359 (0.261)
  BCVA final | 0.353 (0.320)

5. Primary Outcome: Conjunctival Redness
Description: The Efron Grading Scales for Contact Lens Complications includes a standardized method for quantifying the level of conjunctival redness noted on slit lamp examination. The scale ranges, in whole numbers, from 0 to 4, with 0 indicating that conjunctival redness is not present (better outcome) and 4 indicating that the most severe redness is present (worse outcome).
Time Frame: baseline and one month post treatment initiation
Population: All subjects who completed study
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 9
Number analyzed (eyes) | 18
score on a scale
  Conjunctival redness (modified Efron scale) at baseline | 16.78 (8.11)
  Conjunctival redness (modified Efron scale) at 1 month post treatment initiation | 10.2 (7.21)

6. Primary Outcome: Tolerability Questionnaire Score
Description: Subjects completed questionnaires regarding PROSE device comfort and fit (Tolerability Questionnaire, scale 0 to 10, higher score means better outcome), measured pre and post initiation of 0.05% cyclosporine treatment. Total tolerability score is a composite score sum of SIX questions (maximum score of 60).
Time Frame: baseline and one month post initiation treatment
Population: Subjects who completed the study
Measure: Mean (Standard Deviation); unit: tolerability score
Arm/Group | Single Arm
Number analyzed (Participants) | 9
tolerability score
  Total tolerability questionnaire score at baseline | 46.22 (11.40)
  Total tolerability questionnaire score 1 month post initiation of treatment | 47.56 (11.22)

7. Primary Outcome: Automated Conjunctival Redness Without PROSE Device on the Eye
Description: Conjunctival redness score measured using the automated imaging system Keratograph 5M R-Scan. The Keratograph 5M R-scan is an imaging device which classifies bulbar and limbal conjunctival redness. The R-Scan detects blood vessels in the conjunctiva and evaluates the degree of redness. The minimum score per eye is 0 (no redness present, better outcome), while the maximum score per eye is 4 (most severe redness present, worse outcome).
Time Frame: baseline and one month post treatment initiation
Population: Sixteen of the eighteen study eyes (8 participants) had adequate K5MRS image acquisition for analysis. Image acquisition was not obtained (machine unable to acquire) for several conjunctival sections at several time points for one subject, so this subject was excluded from the K5MRS analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 8
Number analyzed (eyes) | 16
score on a scale
  Conjunctival redness (K5MRS score) at baseline | 3.74 (1.09)
  Conjunctival redness (K5MRS score) 1 month post initiation of treatment | 3.25 (1.00)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Arm One: One subject withdrew from the study for ocular burning and stinging.
Arm/Group | Arm One
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm One (N=10)
ocular burning and stinging (Eye disorders) | 1 (1) — Subject experienced ocular burning and stinging
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm One (N=10)
ocular burning and stinging (Eye disorders) | 1 (1) — One subject experienced ocular burning and stinging and was withdrawn from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT04918823/Prot_002.pdf
  • Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT04918823/SAP_003.pdf